CLINICAL TRIAL: NCT01555320
Title: Clinical Assessment of Complementary Treatment With Qishen Yiqi Dripping Pills on Ischemic Heart Failure (CACT-IHF) A Randomized, Double-blind, Multicenter, Placebo-controlled Trial
Brief Title: Clinical Assessment of Complementary Treatment With Qishen Yiqi Dripping Pills on Ischemic Heart Failure
Acronym: CACT-IHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government)
Responsible Party: Principal Investigator, Jingyuan Mao, Prof., First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201007001-02
Record Dates: First submitted 2012-02-29; First posted 2012-03-15 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Ischemic Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qishen Yiqi dripping pills dummy (Placebo Comparator)
  Interventions: Drug: Qishen Yiqi dripping pills dummy
- Qishen Yiqi Dripping Pills (Experimental)
  Interventions: Drug: Qishen Yiqi Dripping Pills

INTERVENTIONS:
Drug: Qishen Yiqi Dripping Pills — One packet of Qishen Yiqi Dripping Pills (0.52g) will be given three times a day in addition to regular western medications for the first 6 months, and regular western medications only for the subsequent 6 months.
  Arms: Qishen Yiqi Dripping Pills
Drug: Qishen Yiqi dripping pills dummy — One packet of Qishen Yiqi Dripping Pills dummy (0.52g) will be given three times a day in addition to regular western medications for the first 6 months, and regular western medications only for the subsequent 6 months.
  Arms: Qishen Yiqi dripping pills dummy

SUMMARY:
CACT-IHF aims to evaluate the clinical efficacy and safety of Qishen Yiqi Dripping Pills in treating ischemic heart failure. Meeting the diagnosis, inclusion and exclusion criteria, the study plans to recruit 640 cases from 35 upper class hospitals in China, who are divided into two groups (treatment and control group) by central randomization service. The treatment group will be administrated with one bag of Qishen Yiqi Dripping Pills (0.52g/bag) three times a day in addition to standardized western medications. Whereas the control group will be given one bag of Qishen Yiqi Dripping Pills dummy (0.52g/bag) three times a day in addition to standardized western medications. Efficacy indicators include primary indicator (6 minute walk test) and secondary indicators: composite endpoint consisting of all-cause death, emergency/re-admission to hospital due to HF, frequency of re-admission due to cardiovascular disease, acute coronary syndrome, severe arrhythmia, cardiac shock, revascularization, stroke, pulmonary embolism and peripheral vascular incidences, etc.; Brain Natriuretic Peptide; echocardiography; cardiothoracic ratio; NYHA cardiac function classification; Minnesota life quality scale; scores from the four traditional chinese medicine (TCM) diagnostic methods). Other indicators include blood cholesterol, triglyceride, high density cholesterol and low density cholesterol. Safety indicators include blood pressure, heart rate, blood and urine routine tests, liver and renal function tests, serum electrolytes, electrocardiogram and adverse events. All of the patients will receive interventional drug treatment for 6 months. Follow up is needed on the 1st, 3rd, 6th, 9th, 12th month after recruitment. All patients will be followed up until the end of study (Refers to the 12th month of the last case recruited into the study).

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 79
* Patients with ischemic heart failure：

  * LVEF less than or equal to 45% measured by echocardiography in modified Simpson method
  * History of prior myocardial infarction with or without percutaneous coronary intervention (PCI) or/and coronary artery bypass grafting (CABG);
  * Coronary angiography (CAG) or coronary CTA shows more than or equal to 50% stenosis in at least one of the main coronary arteries with or without revascularization, of which the researcher thinks that it is closely related to heart failure;
  * With or without dyspnea, fatigue and fluid retention (edema) etc.
* History of heart failure or present with heart failure symptoms for at least 3 months;
* New York Heart Association (NYHA) Class II to IV;
* Submitted informed consent

Exclusion Criteria:

* Acute heart failure or acute exacerbation of chronic heart failure
* Those who have one of the following diseases:

  * Acute coronary syndrome within 30 days
  * Revascularization therapy within 6 months
  * Uncontrolled hypertension with systolic pressure more than or equal to 180mmHg and/or diastolic pressure more than or equal to 110mmHg
  * Second degree type 2 or worse sinoatrial/atrioventricular block without implantation of pacemaker or uncontrolled malignant cardiac arrhythmia
  * Dilated cardiomyopathy
  * Hypertrophic obstructive cardiomyopathy
  * Myocarditis
  * Pulmonary artery embolism
  * Severe valvular heart disease
  * Pulmonary heart disease
  * Stroke within 6 months
* Cardiac resynchronization therapy
* Applied diuretics, cardiotonic agents or vasodilators intravenously within 7 days
* Severe endocrine diseases such as hyperthyroidism, etc.
* History of malignant tumor
* Hemoglobin (HB )≤ 9g/dl
* Alanine aminotransferase (ALT) > 2 times the upper limit of normal
* Serum creatinine > 265 μmol/L
* Mental disorder
* Being pregnant, planning for pregnancy or breastfeeding
* Suspicious or definite allergy to intervention drugs
* Participated in other trials within 2 months
* Unable to walk autonomously due to physical disabilities

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
6MWT distance | 0 month
6MWT | 3rd month
6MWT | 6th month

SECONDARY OUTCOMES:
Composite endpoint | 1st,3rd,6th,9th,12th month
  all-cause death, frequency of emergency/re-admission to hospital due to HF, frequency of re-admission due to cardiovascular disease, acute coronary syndrome, severe arrhythmia, cardiac shock, revascularization, stroke, pulmonary embolism and peripheral vascular incidences, etc.
Brain natriuretic peptide (BNP) | 0,6th month
Echocardiography | 0,6th month
Cardiothoracic Ratio(CR) | 0,6th month
Cardiac function classification, NYHA | 0,1st,3rd,6th,9th,12th month
Minnesota life quality scale | 0,1st,3rd,6th,9th,12th month
Scores from the four TCM diagnostic methods | 0,1st,3rd,6th,9th,12th month
blood and urine routine tests,liver and renal function tests,serum electrolytes,electrocardiogram (ECG) | 0,3rd,6thmonth

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Mao, Dr., Principal Investigator — First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Locations (33):
- China (33):
  - Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Fuwai Hospital, Beijing, Beijing Municipality
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Guangdong Provincial Hospital of TCM, Guangdong, Guangdong
  - Second Affiliated Hospital of TCM College Guiyang, Guiyang, Guizhou
  - 252 Hospital of Chinese People's Liberation Army, Baoding, Hebei
  - The 1st Affiliated Hospital of Heilongjiang Traditional Chinese Medicine University, Heilongjiang, Heilongjiang
  - The First Affiliated Hospital of Henan University of TCM, Zhengzhou, Henan
  - The Affiliated Nanhua Hospital of Nanhua University, Hengyang, Hunan
  - Jiangsu Province Traditional Chinese Medicine Hospital, Nanjing, Jiangsu
  - Nanjing Hospital of T.C.M, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangxi University of TCM, Nanchang, Jiangxi
  - The Affiliated Hospital To Changchun University of Chinese Medicine, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - Shandong Province Traditional Chinese Medicine University Affiliated Hospital, Shandong, Shandong
  - Ruijin Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Shanghai, Shanghai Municipality
  - Shanghai Shuguang Hospital, Shanghai, Shanghai Municipality
  - Traditional Chinese Medicine Hospital of Shan Xi Province, Taiyuan, Shanxi
  - Teaching Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - Affiliated Hospital of Medical College of Chinese People's Armed Police Forces, Tianjin, Tianjin Municipality
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Second Affiliated Hospital of Tianjin University of TCM, Tianjin, Tianjin Municipality
  - The 2nd Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tian Jin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Academy of Traditional Chinese Medicine Affliated Hospital, Tianjin, Tianjin Municipality
  - Traditional Chinese Medical Hospital of Xinjiang Uyghur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Anhui University of TCM, Anhui
  - Dong Fang Hospital, Beijing

REFERENCES:
- [Derived] Zhou Z, Wang S, Du Y, Zhao Z, Bi Y, Su Q, Hou Y, Wang X, Mao J. Effect of Qishen Yiqi Dripping Pill on Clinical Outcomes in Patients with Ischemic Heart Failure: A Post-Hoc Analysis of the CACT-IHF Randomized Trial. Drug Des Devel Ther. 2025 Nov 15;19:10163-10174. doi: 10.2147/DDDT.S556373. eCollection 2025. PMID 41268060
- [Derived] Hou YZ, Wang S, Zhao ZQ, Wang XL, Li B, Soh SB, Mao JY. Clinical assessment of complementary treatment with Qishen Yiqi dripping pills on ischemic heart failure: study protocol for a randomized, double-blind, multicenter, placebo-controlled trial (CACT-IHF). Trials. 2013 May 14;14:138. doi: 10.1186/1745-6215-14-138. PMID 23672353